CLINICAL TRIAL: NCT06208852
Title: The Social Media-Based Parenting Program for Women With Postpartum Depressive Symptoms: Virtual Patient Navigation During a Pandemic
Brief Title: Virtual Patient Navigation During a Pandemic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 19-016174-B; R61MH118405 (NIH); 19-016174 (Other: CHOP)
Record Dates: First submitted 2023-12-21; First posted 2024-01-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Post-partum Depression
Keywords: post-partum depression; mental health; child and maternal health; patient navigator
MeSH Terms: conditions — Depression, Postpartum; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The sub-study will involve a rigorous mixed-methods design. The qualitative phase of the sub-study will consist of semi-structured interviews. During the semi-structured interviews, 10 eligible women will be recruited to identify barriers and facilitators to accessing virtual mental health services. This information will be used to adapt an evidence-based patient navigation intervention for virtual use. For the intervention phase of the sub-study, 30 women with persistent postpartum depression (PPD) symptoms will be recruited to participate in the adapted virtual navigator program using rapid cycle testing over a 2-month period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qualitative phase (No Intervention): The qualitative phase of the sub-study will consist of semi-structured interviews. During the semi-structured interviews, 10 eligible women will be recruited to identify barriers and facilitators to accessing virtual mental health services during the pandemic. This information will be used to adapt an evidence-based patient navigation intervention for virtual use.
- Intervention Phase (Experimental): For the intervention phase of the sub-study, 30 women with persistent postpartum depression symptoms will be recruited to participate in the adapted virtual navigator program using rapid cycle testing over a 2-month period.
  Interventions: Other: Virtual Navigator Program

INTERVENTIONS:
Other: Virtual Navigator Program — For the intervention phase of the sub-study, 30 women with persistent PPD symptoms will be recruited to participate in the adapted virtual navigator program using rapid cycle testing over a 2-month period. These women will be enrolled and consented to receive virtual patient navigation for 2 months. Investigators will conduct rapid cycle testing in which we will evaluate satisfaction, feasibility, and target engagement of the intervention after every 10 participants in order to make rapid cycle changes prior to enrolling the next 10 participants. Women will communicate virtually with the PN by means of telephone, text messaging, Facetime, or other virtual modality of their choice. The Primary Navigator (PN) will meet with families at the beginning of the study to review results of depression screens and community mental health (MH) resources. The PN will partner with participants, engage them in the program, and provide ongoing communication with participants and MH clinicians.
  Arms: Intervention Phase

SUMMARY:
The sub-study will involve a rigorous mixed-methods design. The qualitative phase of the sub-study will consist of semi-structured interviews. During the semi-structured interviews, 10 eligible women will be recruited to identify barriers and facilitators to accessing virtual mental health services. This information will be used to adapt an evidence-based patient navigation intervention for virtual use. For the intervention phase of the sub-study, 30 women with persistent postpartum depression symptoms will be recruited to participate in the adapted virtual navigator program using rapid cycle testing over a 2-month period.

DETAILED DESCRIPTION:
In the qualitative phase of the sub-study, 10 participants who are either former participants from the R61 Phase (IRB 19-016174) of the Main Randomized Clinical Trial (RCT), or have been referred, are actively enrolled, or withdrawn in the R33 Phase (IRB 22-019784) of the Main RCT, will be recruited to participate in semi-structured interviews. In the intervention phase of the sub-study, 30 eligible women who are either former participants from the R61 Phase (IRB 19-016174) of the Main RCT, or have been referred, enrolled but completed participation, or withdrawn from the R33 Phase (IRB 22-019784) of the Main RCT, but not actively engaged with mental health services, will be enrolled and consented to receive virtual patient navigation for 2 months. The qualitative phase will involve audio-recorded semi-structured interviews to identify barriers and facilitators to virtual and in-person mental health services. These interviews will then inform the intervention phase which involves the adaptation of an existing mental health navigation intervention for a virtual environment. For both phases of the sub-study, those who agree to participate will be asked to verbally agree to the approved HIPAA form and sign the informed consent form.

For the qualitative phase of the sub-study, 10 eligible women will participate in a 30-40 minute semi-structured interview. Following written informed consent, the participating mother will then participate in a 30-40 minute semi-structured interview. The interview will consist of questions regarding barriers and facilitators to accessing mental health services during a pandemic. The interviews will be audiotaped and transcribed. In the event that the interview cannot be completed in person, a research staff member will complete the interview over the phone with the participant. Transcripts of interviews will be reviewed by 2-3 investigators. Transcripts will be coded and emergent themes related to barriers and facilitators to virtual navigation will be identified using inductive means. Initial codes will be developed inductively through consensus of the investigative team. Themes pertaining to child and family factors and benefits and barriers to mental health service use in a virtual environment will be identified. Investigators will use NVivo, a qualitative software program, to facilitate coding of transcripts and identification of themes. This information will be used to adapt an evidence-based patient navigation intervention for virtual use.

For the intervention phase of the sub-study, 30 women with persistent postpartum depression symptoms will be recruited to participate in the adapted virtual navigator program using rapid cycle testing over a 2-month period. These women will be enrolled and consented to receive virtual patient navigation for 2 months. Investigators will conduct rapid cycle testing in which the investigators will evaluate satisfaction, feasibility, and target engagement of the intervention after every 10 participants in order to make rapid cycle changes prior to enrolling the next 10 participants.

Women will communicate virtually with the patient navigator by means of telephone, text messaging, Facetime, or other virtual modality of their choice. The patient navigator will meet with families at the beginning of the study to review results of depression screens and community mental health resources. The patient navigator will partner with participants, engage them in the program, and provide ongoing communication with participants and mental health clinicians. The patient navigator will contact participants weekly by phone, text messaging, email, or any other modality depending on participant preference to monitor initiation and completion of referral, identify concerns and/or barriers to referral completion, and assist participants with problem-solving to identify potential barriers and solutions to complete mental health referrals. Specific barriers and proposed solutions will be identified in the qualitative study above. Using virtual means, the patient navigator will also communicate with mental health clinicians to clarify appointments and address emerging issues. A fidelity checklist will be adapted to assess self-reported task completion by the patient navigator.

All participants will be monitored monthly for depressive symptoms and suicidality. Those who report worsening depressive symptoms (EPDS>20) or suicidality (affirmative response to Question #10 on the EPDS) will be contacted immediately by study staff and an existing suicide protocol from the parent study will be initiated.

ELIGIBILITY:
Inclusion Criteria

Qualitative Phase:

Women who:

1. Are either former participants from the R61 Phase (IRB 19-016174) of the Main RCT, or have been referred, are actively enrolled, or withdrawn from the R33 Phase (IRB 22-019784) of the Main RCT.
2. Are > 18 years of age
3. Speak and read in English
4. Have access to a smart phone or computer tablet with internet access
5. Have an infant < 12 months of age

Intervention Phase:

Women who:

1. Are not actively engaged with MH services
2. Screen positive for postpartum depression (score>9) on the EPDS
3. Are > 18 years of age
4. Speak and read in English
5. Have access to a cellular phone with texting capabilities

Exclusion Criteria

Qualitative Phase:

Women who:

1. Report suicidality (i.e., suicidal ideation and/or behavior) on the EPDS (Question #10) at enrollment.
2. Report severe depressive symptoms (EPDS>20) at enrollment.
3. Have a substantiated report of child maltreatment

Children who:

1. Were born premature (estimated gestational age<35 weeks)
2. Have been diagnosed with congenital malformations or genetic syndromes which place them at risk of developmental delays
3. Are already currently receiving early intervention services for developmental delays at baseline

Intervention Phase:

Women who:

1. Report suicidality (i.e., suicidal ideation and/or behavior) on the EPDS (Question #10) with a response of "sometimes," or "yes, quite often" at participating pediatric practice
2. Report suicidality (i,e, suicidal ideation and/or behavior) on the EPDS (Question #10) and also endorse any of the follow up questions at a participating pediatric practice:

   i. Have you ever felt that life is not worth living? ii. Has this feeling occurred in the past week? iii. Have you ever wanted to kill yourself? iv. Did you ever make a plan to kill yourself? v. Have you ever attempted suicide?
3. Have a substantiated report of child maltreatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Birth-mothers who experienced PPD symptoms
Enrollment: 40 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Qualitative: Barriers and facilitators to virtual and in-person mental health services | Baseline
  the main objective is to identify barriers and facilitators to virtual and in-person mental health services in order to adapt a patient navigation intervention for virtual use.
Intervention: Target engagement of the Patient Navigator | Baseline, 2 months.
  To determine target engagement of the virtual PN, changes in the The Barriers to Mental Health Services Scale Revised (BMHSS-R ) measured at baseline and at the 2-month follow-up visit will be assessed.
Intervention: Feasibility | Baseline, 2 months
  To assess the feasibility of the intervention, the proportion of eligible women who enroll and complete the study will be examined.
Intervention: Acceptability | 2 months
  To assess acceptability, participants will complete a measure of satisfaction that will include a closed question assessing their satisfaction with the virtual PN using a 5-point likert-scaled response category and an open-ended question concerning their likes and dislikes.

SECONDARY OUTCOMES:
Intervention: Changes in depressive symptoms | Baseline, 1month, 2 months
  The EPDS is a validated 10-item self-report measure of depressive symptoms with strong evidence for reliability, validity, and utility in varying populations. It has been used extensively in mental health research and provides cutpoints to determine the severity of depressive symptoms. It includes a question on suicidal thoughts and wishes (#10) that will be used to monitor for suicidality. The total score will be used with scores of 10 or higher representing minor or moderate depression and scores of 20 or greater representing severe depression.
Intervention: Mental health treatment usage | Baseline, 1 month, 2 months
  Outside mental health treatment will be measured monthly using the item from the National Comorbidity Survey (NCS) concerning any mental health service use.

CONTACTS AND LOCATIONS:
Overall Officials: James Guevara, MD, MPH, Principal Investigator — Children's Hospital of Philadelphia; Rhonda Boyd, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete, cleaned, and de-identified dataset will be made available to other investigators after all analyses have been conducted and within twelve months of the end of the final year of funding to allow for publication of all study aims. To obtain this data set, other investigators will need to contact the study Principal Investigator (PI) who will provide a data sharing agreement. The data sharing agreement will permit a deidentified data set to be shared once an Institutional Review Board (IRB) protocol has been approved at the investigators' home institution and the investigators have signed a pledge to not attempt to identify individual study subjects. The data set will be made available on a Compact Disc Read-Only Memory (CD-ROM) or through a secure File Transfer Protocol (FTP) site.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after the end of the final year of funding.

REFERENCES:
- [Background] Guevara JP, Morales K, Mandell D, Mogul M, Charidah T, Luethke M, Min J, Clark R, Betancourt L, Boyd R. Social Media-based Parenting Program for Women With Postpartum Depressive Symptoms: An RCT. Pediatrics. 2023 Mar 1;151(3):e2022058719. doi: 10.1542/peds.2022-058719. PMID 36808207